CLINICAL TRIAL: NCT06303752
Title: Repairing Peri-Anal Fistulas With Regenerative Cell Therapeutics
Brief Title: Tissue Therapy of Transsphincteric Anal Fistula
Acronym: REP-PAF
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Karam Matlub Sørensen, PhD, Primary Investigator (PI), University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 260-2021-NQ; 2022-502659-73 (EudraCT Number)
Record Dates: First submitted 2024-02-25; First posted 2024-03-12 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Anal Fistula
Keywords: anal fistula; stem cells; ADRC
MeSH Terms: conditions — Rectal Fistula | interventions — Lipectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Autologous ADRC (Experimental): Allocated patients will be treated for the fistula by combined surgical debridement of the fistula tract, closure of the internal orifice and injection of 30 ml lipoaspirate around the entire length of the fistula tract. Lipoaspirate will be harvested from the anterior abdominal wall under the same operation. Two hours later, the patient will receive injection of 5 ml suspension including 30 million autologous adipose-derived regenerative cells ADRC and injected at the same site of the lipoaspirate injection.
  Interventions: Drug: ADRC injection
- allogenic ADRC001 (Experimental): Allocated patients will be treated for the fistula by combined surgical debridement of the fistula tract, closure of the internal orifice and injection of 30 ml lipoaspirate around the entire length of the fistula tract. Lipoaspirate will be harvested from the anterior abdominal wall under the same operation. Two hours later, the patient will receive injection of 5 ml suspension including 30 million cultured allogenic adipose-derived regenerative cells ADRC001 and injected at the same site of the lipoaspirate injection.
  Interventions: Drug: ADRC001 injection

INTERVENTIONS:
Drug: ADRC injection — Allocated patients will receive injection of 5 ml suspension including 30 million autologous adipose-derived regenerative cells ADRC and injected at the same site of the lipoaspirate injection.
  Other Names: Liposuction; Surgical debridement of fistula tract and closure of internal orifice; Injection of lipoaspirate
  Arms: Autologous ADRC
Drug: ADRC001 injection — Allocated patients will receive injection of 5 ml suspension including 30 million allogenic adipose-derived regenerative cells ADRC001 and injected at the same site of the lipoaspirate injection.
  Other Names: Liposuction; Surgical debridement of fistula tract and closure of internal orifice; Injection of lipoaspirate
  Arms: allogenic ADRC001

SUMMARY:
This clinical study aims to evaluate the outcome of the treatment of complex perianal fistulas (PAF) by the combination of minimal surgical debridement with regenerative cellular therapeutics.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo screening serology and preoperative work-up to determine eligibility for study entery. Patients who meet the eligibility requirements will be treated for their fistulas by combined minor surgical debridement of the fistula tract and closure of the internal orifice as well as liposuction from the abdominal wall. Regenerative cells- enriched lipoaspirate will be injected around the entire length of the fistula tract. The first five patients will receive their own regenerative cells and act as donors for the next included patients, but they will not be included in the final analysis. The rest of the included patients (70) will be randomized in double-blinded manner (participant and investigator) in a 1:1 ratio to either recieve own regenerative cells (ADRC Adipose-Derived Regeneative Cells) or donated cultured regenerative cells (ADRC001). All included patients will be scheduled for follow-up at 3, 6 and 12 months after treatment.

ELIGIBILITY:
Inclusion criterion:

Adult patients (>= 18years) with complex anal fistula (high transsphincteric or suprasphincteric), with involvement of more 30% of the anal sphincter referred to the surgical department at Odense University Hospital for treatment, and who are:

* able to communicate with Danish language
* able to provide informed consent
* having address in the region of southern Denmark during the study

Exclusion criteria:

1. Signs of suppuration/cavitation around the fistula
2. Simple or low anal fistula, which can be treated by simple surgical incision
3. Ano-vaginal and recto-vaginal fistula
4. The presence of more than one fistula tract, more than two external orifices or more than one internal orifice
5. Inflammatory Bowel Disease
6. Immunosuppression (due to clinical condition or medical therapy)
7. Malignancy within 5 years
8. Previous radiotherapy of the abdomen and pelvis
9. BMI under 18.5
10. Allergy against the antibiotics: Penicillin and streptomycin.
11. Coagulopathy
12. Pregnancy and lactation (positive HCG (human chorionic gonadotropin) test)
13. Verified syphilis, HIV, or hepatitis on screening test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2027-10-08 (Estimated); Study Completion 2028-10-08 (Estimated)

PRIMARY OUTCOMES:
Healing rate (percentage) | at 6 and 12 months follow-up
  Clinical healing is defined as closure of the external opening(s), absence/cessation of discharge and swelling by palpation.

SECONDARY OUTCOMES:
QoL | at12 months follow-up.
  functional outcome regarding quality of life, measured by Short Form SF-36 Rand questionnaire.
Fecal Incontinence | at12 months follow-up.
  functional outcome regarding fecal incontinence, measured by Wexner Fecal Incontinence score.
Risk factors for recurrence of fistula. | at12 months follow-up.
  Risk factors for recurrence of fistula including demography, prevoius surgery for fistula, disease duration and treatment arm.
Radiological healing. | at12 months follow-up.
  Radiological healing, defined as no visible fistula or fluid collection more than 5 mm at MR imaging.
Treatment efficacy. | at12 months follow-up.
  comparison of the healing rate of the fistula between patients receiving ADRC and patients receiving ADRC001 (autologous vs. allogenic cells)
Cellular composition | at 3 months follow-up.
  Definition of the cellular compisition of the ADRC and ADRC001 regarding cellular surface markers (CD14, CD31, CD34, CD45, CD73, CD90, CD105, CD235a, HLA-ABC og HLA-DR) using flowcytometry.
Transplantation-related alloantibodies | at12 months follow-up.
  Registration of the number of patients developing serum alloantibodies specific to donor genotypes, by assessment of anti-HLA (class I and II).

CONTACTS AND LOCATIONS:
Overall Officials: Karam M Sørensen, Principal Investigator — OUH
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No